CLINICAL TRIAL: NCT05286346
Title: A Multi-Center, Randomized, Open-label, Parallel, Active-controlled, Non-inferiority, Phase IV Clinical Trial to Evaluate the Safety and Efficacy of Switching to Tenolid Tab (Tenofovir Disoproxil) From Viread Tab (Tenofovir Disoproxil Fumarate) in Chronic Hepatitis B Patients on Treatment With Tenofovir Disoproxil Fumarate
Brief Title: Clinical Study to Evaluate the Safety and Efficacy of Switching to Tenofovir Disoproxil From Tenofovir Disoproxil Fumarate in Patients With Chronic Hepatitis B
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samjin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TNLD02
Record Dates: First submitted 2022-02-25; First posted 2022-03-18 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Tenolid Tab
  Interventions: Drug: Tenofovir disoproxil 245mg
- Control group (Active Comparator): Viread Tab
  Interventions: Drug: Tenofovir disoproxil fumarate 300mg

INTERVENTIONS:
Drug: Tenofovir disoproxil 245mg — 1 tablet q.d. for 48 weeks
  Arms: Experimental group
Drug: Tenofovir disoproxil fumarate 300mg — 1 tablet q.d. for 48 weeks
  Arms: Control group

SUMMARY:
This is a Phase4, multicenter, open-label, randomized study to demonstrate that the Tenolid Tab switching group is non-inferior to the virologic suppression effect compared to the Viread Tab continuous administration group and evaluate the safety of Tenolid Tab. This clinical trial was conducted on patients who were taking Viread Tab as monotherapy for more than 48 weeks for chronic hepatitis B.

At the time of screening(Visit 1), information on factors related to medical history and prognosis including Viread Tab administration were collected retrospectively from the subjects who voluntarily signed the informed consent form (ICF). Only subjects who are determined to be suitable for the study eligibility(inclusion/exclusion) criteria as a result of the screening evaluations are randomized in a 1:1 ratio to one of the two groups at the baseline.

Subjects will receive investigational product start on the next day of randomization for 48 weeks. Subjects will visit to the study site on 12, 24, 36, 24 weeks after starting dosing investigational product and evaluated for effectiveness of virologic suppression and safety.

ELIGIBILITY:
Inclusion Criteria:

1. As of the date of written consent, adults aged 19 or above
2. Patients with chronic hepatitis B
3. For chronic hepatitis B, Viread Tab. monotherapy† for more than 48 weeks, HBV suppression‡(virologic suppression) was confirmed, and it was determined that Tenofovir monotherapy for more than 48 weeks would be required.

   † However, patients who take Viread Tab for more than 48 weeks before screening but do not take Viread Tab at the time of screening and discontinue the administration within 4 weeks until the time of randomization can be registered. (treatment gap ≤ 28 days)
   * HBV DNA < 400 copies/mL (=69 IU/mL*) * IU/mL is converting to copies/mL by unit for each institution. (Ex: 5.8 copies/mL = 1 IU/mL)
4. Subject who voluntarily consents to participate in the clinical trial and signs an informed consent

Exclusion Criteria:

1. Patients with liver cancer or decompensated liver cirrhosis* *Cirrhosis with clinical signs/symptoms of decompensation (jaundice, ascites, variceal bleeding, hepatic coma)
2. Patients with Hepatitis C virus (HCV), human immunodeficiency virus (HIV) with overlapping infections (HCV Ab positive, HIV Ab positive) However, if the HCV Ab or HIV Ab test result is judged to be 'false positive' by the investigator, HCV or HIV infection can be confirmed through additional confirmatory tests (HCV, HIV RNA test), etc.
3. Patients with other clinically significant liver disease (Hemochromatosis, Wilson's disease, Alcoholic liver disease, Autoimmune hepatitis, α-1 antitrypsin deficiency)
4. Patients confirmed by laboratory test results as followings

   * Severe anemia: Hemoglobin < 8g/dL ② Inadequate renal function: eGFR (Ccr, Cockcroft-Gault formula) < 50 mL/min ③ Inadequate hepatic function:

     * Total bilirubin > 3.0 mg/dL
     * Albumin < 2.8 mg/dL
     * Prothrombin Time(PT) > INR 2.2
5. Patients with malignant tumors diagnosed within 5 years prior to screening However, in the case of basal cell carcinoma or squamouscell carcinoma of the skin, it is possible to participate in the clinical trial if it is judged to be 'cured' at the discretion of the investigator after surgery (treatment),.
6. Patients who are scheduled for an organ transplantation or who have undergone organ transplantation surgery
7. Patients with a history of clinically significant neuropsychiatric disorders, alcoholism, or drug dependence
8. Patients known to have hypersensitivity or allergy to components of investigational products or similar drugs
9. Patients who administered immunosuppressive drugs within 24 weeks prior to screening or who administered systemic corticosteroids over a limited dose (equivalent to prednisolone 10 mg/day) for 4 consecutive weeks or more.
10. Patients who are expected to require administration of the following drugs during the clinical trial period

    ① Immunosuppressive drug

    ② Systemic corticosteroids above a limited dose (equivalent to prednisolone 10 mg/day) for 2 consecutive weeks or more

    ③ Drugs affecting renal excretion, drugs inducing nephrotoxicity or hepatotoxicity

    ④ Anti-HBV drugs other than Tenofovir (ex. emtricitabine, lamivudine, telbivudine, clevudine, entecavir, interferone)

    ⑤ Patients who administered hepatotonics at a stable dose for more than 3 months before screening can be registered.
11. Those who have a history of fractures requiring bone mineral density (BMD) monitoring or are at risk of osteopenia, who are judged unable to participate in clinical trials according to the investigator's judgment
12. For pregnant, lactating and reproductive women, patients who do not consent to contraception by a medically accepted method (surgical sterilization, intrauterine device, condom or diaphragm) during the clinical trial period
13. Patients who participated in another clinical trial within 12 weeks prior to screening and received investigational drugs or investigational devices.
14. In addition to the above, subject considered ineligible to participate in this study by the investigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2020-08-10 (Actual)

PRIMARY OUTCOMES:
Inhibiting† rate of HBV virus at 48 weeks after baseline †HBV DNA < 400 copies/mL (=69 IU/mL*) *IU/mL is converting to copies/mL by unit for each institution. (ex: 5.8 copies/mL = 1 IU/mL) | 48 weeks

SECONDARY OUTCOMES:
Inhibiting† rate of HBV virus at 12, 24 and 36 weeks after baseline †HBV DNA < 400 copies/mL (=69 IU/mL*) * IU/mL is converting to copies/mL by unit for each institution. (ex: 5.8 copies/mL = 1 IU/mL) | 12, 24, 36 and 48 weeks
Undetected‡ rate of HBV virus at 12, 24, 36 and 48 weeks after baseline ‡ The lower limit of quantification (LLOQ) for each institution is used, and if it is less than the LLOQ, the HBV DNA level is set to '0'. | 12, 24, 36 and 48 weeks
Change of HBV DNA(log10 copies/mL) at 12, 24, 36 and 48 weeks from baseline | 12, 24, 36 and 48 weeks
Loss rate of HBeAg in HBeAg(+) patients at 12, 24, 36 and 48 weeks after baseline | 12, 24, 36 and 48 weeks
Seroconversion† rate of HBeAg in HBeAg(+) patients at 12, 24, 36 and 48 weeks after baseline †Generation of anti-HBe | 12, 24, 36 and 48 weeks
Loss rate of HBsAg in HBsAg(+) patients at 12, 24, 36 and 48 weeks after baseline ④ Seroconversion† rate of HBsAg in HBsAg(+) patients at 12, 24, 36 and 48 weeks after baseline †Generation of anti-HBs | 12, 24, 36 and 48 weeks
Seroconversion† rate of HBsAg in HBsAg(+) patients at 12, 24, 36 and 48 weeks after baseline †Generation of anti-HBs | 12, 24, 36 and 48 weeks
Normal rate of ALT at 12, 24, 36 and 48 weeks after baseline | 12, 24, 36 and 48 weeks
Change of ALT at 12, 24, 36 and 48 weeks from baseline | 12, 24, 36 and 48 weeks
Virologic breakthrough* rate within 48 weeks after baseline *HBV DNA ≥ 400 copies/mL: twice in a row at intervals of 2 weeks or more or HBV DNA levels: increasing by 1log10 from Nadir levels of each subject twice in a row (HBV DNA <400 copies/mL) | 12, 24, 36 and 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Seong Uk Lee, Principal Investigator — Dong-A University Hospital
Locations (1):
- Dong-A University Hospital, Busan, South Korea